CLINICAL TRIAL: NCT05796375
Title: Replacing Invasive Cystoscopy With Urine Testing for Non-muscle Invasive Bladder Cancer Surveillance
Acronym: ReplaceCysto
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: White River Junction Veterans Affairs Medical Center (U.S. Federal Agency)
Collaborators: National Cancer Institute (NCI) (NIH); University of Texas Southwestern Medical Center (Other); Medical University of South Carolina (Other)
Responsible Party: Principal Investigator, Florian Schroeck, Chief, Section of Urology, White River Junction Veterans Affairs Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 1732756; R37CA275916 (NIH); 1R37CA275916-01 (NIH)
Record Dates: First submitted 2023-03-21; First posted 2023-04-03 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Non-muscle-invasive Bladder Cancer
Keywords: Bladder; Cancer; Urology; Cystoscopy; Xpert; EpiCheck; Urine test
MeSH Terms: conditions — Non-Muscle Invasive Bladder Neoplasms; Neoplasms | interventions — Cystoscopy

STUDY DESIGN:
Intervention Model Description: Health care delivery parallel trial with 1:1:1 randomization
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (3):
- Frequent Cystoscopy (Active Comparator): Cystoscopy is conducted at 6, 12, 18, and 24 months for patients undergoing surveillance for low grade intermediate-risk non-muscle invasive bladder cancer
  Interventions: Procedure: Cystoscopy
- Xpert Urine Test (Experimental): Xpert arm includes urine testing using the Xpert Bladder Cancer Monitor urine test at 6 and 18 months. Cystoscopy is conducted at 12 and 24 months for patients undergoing surveillance for low grade intermediate-risk non-muscle invasive bladder cancer
  Interventions: Procedure: Cystoscopy; Diagnostic Test: Xpert Bladder Cancer Monitor urine test
- EpiCheck Urine Text (Experimental): EpiCheck arm includes urine testing using the Bladder EpiCheck urine test at 6 and 18 months. Cystoscopy is conducted at 12 and 24 months for patients undergoing surveillance for low grade intermediate-risk non-muscle invasive bladder cancer.
  Interventions: Procedure: Cystoscopy; Diagnostic Test: Bladder EpiCheck urine test

INTERVENTIONS:
Procedure: Cystoscopy — Cystoscopy entails direct inspection of the bladder via a cystoscope that is inserted into a patient's urethra.
Diagnostic Test: Bladder EpiCheck urine test — The Bladder EpiCheck is a laboratory-developed test for early-stage non-muscle invasive bladder cancer. The Bladder EpiCheck test is a DNA methylation test that is run on DNA extracted from cell pellet from centrifuged urine according to Standardized Operating Procedures. The test has internal controls and a dedicated software to ensure required quality assurance processes and prompt reporting of results.
  Arms: EpiCheck Urine Text
Diagnostic Test: Xpert Bladder Cancer Monitor urine test — A 4.5 ml sample of voided urine is added to Xpert® Urine Transport Reagent, mixed, and then 4ml of treated urine are transferred to the Sample Chamber of the cartridge. In the cartridge, cells in the urine sample are captured on a filter and lysed by sonication. The released nucleic acid is eluted, mixed with dry RT-PCR reagents, and the solution is transferred to the reaction tube for RT-PCR and detection.
  Arms: Xpert Urine Test

SUMMARY:
The purpose of this research is to determine whether bladder cancer monitoring can be improved by replacing some cystoscopy procedures with urine testing. Specifically, this study examines whether there are any differences in urinary symptoms, discomfort, number of invasive procedures, anxiety, complications, cancer recurrence or cancer progression when some cystoscopy procedures are replaced with urine testing.

DETAILED DESCRIPTION:
This is a multi-site randomized phase 2 trial including 240 patients with early-stage bladder cancer, in which patients will be randomized 1:1:1 to programmatic surveillance with the Xpert bladder cancer urine test, the Bladder EpiCheck urine test, or frequent cystoscopy. The primary outcome will be urinary quality of life measured 1 to 3 days after surveillance.

This study will have three groups, also called "arms": (1) Frequent Cystoscopy Arm, (2) Xpert Urine Test Arm, and (3) Epicheck Urine Test Arm. The aim of Frequent Cystoscopy is to detect any cancer that might have come back within the bladder by frequently inspecting the bladder. Those in the cystoscopy arm will have a cystoscopy procedure at specified time points for two years. The goal of the Xpert Urine Test arm is to detect any cancer that might have come back within the bladder, while decreasing the number of invasive cystoscopy procedures. Those in the Xpert arm will have a Xpert urine test and a check-up with a medical doctor at 6 months and 18 months, and have a cystoscopy procedure at 12 months and 24 months. The aim of the EpiCheck Urine Test arm is to detect any cancer that might have come back within the bladder, while decreasing the number of invasive cystoscopy procedures. Those in the EpiCheck Urine Test arm will have an Epicheck urine test and a check-up with a medical doctor at 6 months and 18 months and will have a cystoscopy procedure at 12 months and 24 months. The study performance period is 24 months.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18 years or older
2. History of low grade intermediate-risk non-muscle invasive bladder cancer, defined as most recent pathology report showing any of the following:

   * multifocal low grade non-invasive urothelial carcinoma of any size
   * solitary low grade non-invasive urothelial carcinoma greater than 3cm in size
   * recurrent low grade non-invasive urothelial carcinoma
3. Stated willingness to comply with all study procedures and availability for the duration of the study
4. No evidence for recurrence at cystoscopy ≤6 months after most recent tumor resection
5. Ability to consent in English or Spanish

Exclusion Criteria:

1. History of total cystectomy of the bladder.
2. History of urinary diversion (e.g., neo-bladder, colon pouch, or ileal conduit).
3. History of muscle-invasive bladder tumor.
4. Pregnancy or lactation.
5. History of urothelial carcinoma of the ureter or renal pelvis status post endoscopic treatment or with evidence of recurrent upper tract disease (inclusion allowed if status post nephroureterectomy and recurrence free at time of inclusion)
6. Anatomic constraints making cystoscopy impossible (e.g., history of urethrectomy, obliterated urethra secondary to stricture).
7. Inability to provide a voided urine sample.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2023-11-17 (Actual); Primary Completion 2028-11-30 (Estimated); Study Completion 2028-12-30 (Estimated)

PRIMARY OUTCOMES:
Quality of Life Questionnaire-Non-Muscle Invasive Bladder Cancer 24 (EORTC QLQ-NMIBC24) | Assessed at 3, 6, 12, 18, and 24 months.
  Measuring change from baseline. Score range: 0-100. Lower score indicates higher quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Florian R Schroeck, MD, MS, Principal Investigator — White River Junction VA Healthcare System
Locations (8):
- United States (8):
  - West Haven VA Medical Center, West Haven, Connecticut
  - Bay Pines VA Healthcare System, Bay Pines, Florida
  - VA Boston Jamaica Plains Campus, West Roxbury, Massachusetts
  - VA St.Louis Healthcare System, St Louis, Missouri
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - Medical University of South Carolina, Charleston, South Carolina
  - UT Southwestern Medical Center, Dallas, Texas
  - White River Junction Veterans Healthcare System, White River Junction, Vermont

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Koo K, Zubkoff L, Sirovich BE, Goodney PP, Robertson DJ, Seigne JD, Schroeck FR. The Burden of Cystoscopic Bladder Cancer Surveillance: Anxiety, Discomfort, and Patient Preferences for Decision Making. Urology. 2017 Oct;108:122-128. doi: 10.1016/j.urology.2017.07.016. Epub 2017 Jul 21. PMID 28739405
- [Background] Schroeck FR, Lynch KE, Li Z, MacKenzie TA, Han DS, Seigne JD, Robertson DJ, Sirovich B, Goodney PP. The impact of frequent cystoscopy on surgical care and cancer outcomes among patients with low-risk, non-muscle-invasive bladder cancer. Cancer. 2019 Sep 15;125(18):3147-3154. doi: 10.1002/cncr.32185. Epub 2019 May 23. PMID 31120559
- [Background] Schroeck FR, Grubb R, MacKenzie TA, Ould Ismail AA, Jensen L, Tsongalis GJ, Lotan Y. Clinical Trial Protocol for "Replace Cysto": Replacing Invasive Cystoscopy with Urine Testing for Non-muscle-invasive Bladder Cancer Surveillance-A Multicenter, Randomized, Phase 2 Healthcare Delivery Trial Comparing Quality of Life During Cancer Surveillance with Xpert Bladder Cancer Monitor or Bladder EpiCheck Urine Testing Versus Frequent Cystoscopy. Eur Urol Open Sci. 2024 Mar 21;63:19-30. doi: 10.1016/j.euros.2024.02.018. eCollection 2024 May. PMID 38558761